CLINICAL TRIAL: NCT00705003
Title: A Double-Blind, Placebo-Controlled Study of a Combination Product (BCI-024 and BCI-049) in Patients With Major Depressive Disorder (MDD)
Brief Title: Efficacy and Safety Study of a Combination Product [Drug:BCI-024 (Buspirone) and Drug:BCI-049 (Melatonin)] to Treat Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BrainCells Inc. (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Fava, Maurizio MD., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBM-IT-01
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Drug Combination (Experimental): BCI-024: over-encapsulated Buspirone tablet 15 mg at bedtime(QD) and BCI-049: over-encapsulated Melatonin tablet 3 mg QD
  Interventions: Drug: BCI-024: over-encapsulated Buspirone tablet 15 mg QD and BCI-049: over-encapsulated Melatonin tablet 3 mg QD
- BCI-024 (Buspirone) (Active Comparator): BCI-024: over-encapsulated Buspirone 15 mg QD
  Interventions: Drug: BCI-024 (Buspirone)
- Matching placebo (Placebo Comparator): Placebo: 1 capsule QD
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: BCI-024: over-encapsulated Buspirone tablet 15 mg QD and BCI-049: over-encapsulated Melatonin tablet 3 mg QD — BCI-024: over-encapsulated Buspirone tablet 15 mg QD and Drug BCI-049: over-encapsulated Melatonin tablet 3 mg QD taken in combination for 6 weeks
  Other Names: Buspar is the brand name of buspirone.
  Arms: Active Drug Combination
Drug: BCI-024 (Buspirone) — Drug BCI-024 (Buspirone) taken once a day at bedtime for 6 weeks.
  Other Names: Buspar is the brand name of buspirone.
  Arms: BCI-024 (Buspirone)
Drug: Matching placebo — Placebo comparator once a day at bedtime for 6 weeks.
  Arms: Matching placebo

SUMMARY:
The primary objective of this study are to evaluate the synergistic effect of a combination product, consisting of drug BCI-024 (buspirone) and drug BCI-049 (melatonin), in reducing symptoms of depression in patients with Major Depressive Disorder.

The safety and tolerability of the combination product will also be evaluated as measured by adverse events and vital signs.

DETAILED DESCRIPTION:
Approximately 120 adult outpatients meeting the study's inclusion and exclusion criteria will be randomized in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male and female subjects between the ages of 18 to 65 meeting the Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder with a Quick Inventory of Depressive Symptomatology-16 Item Self Report (QIDS-SR16) score of >14 at the Screening and Baseline Visits.
* Female subjects must be on a stable and medically reliable form of birth control, must agree to continue use of this birth control during the study, and must have negative urine pregnancy tests at the Screening Visit.

Exclusion Criteria:

* Subjects with any other psychiatric Axis-I disorder as a principal diagnosis within 6 months of screening or subjects with a history of obsessive compulsive disorder, psychotic disorder, bipolar disorder, or mental retardation at any time are not eligible for the study.
* Subjects who pose a suicidal risk or who have a history of eating disorder or substance dependence within 6 months of screening, or a history of substance abuse within 3 months of screening are also ineligible.
* Subjects with clinically significant abnormalities on any Screening or Baseline assessments, including laboratory tests, are excluded.
* Subjects with a known intolerance to either buspirone or melatonin are excluded, as are subjects with clinically significant medical or psychiatric conditions that might be detrimental to the subject should they participate in the study.
* Subjects who have used selective serotonin reuptake inhibitors (SSRIs) within 2 weeks of Screening (within 4 weeks for fluoxetine) are excluded as are subjects requiring concomitant use of antipsychotic and anxiolytic medications and any drugs with known psychotropic properties. Concomitant medications that are not excluded by the protocol and that are taken chronically must be at a stable dosage for at least 4 weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Andrew A Nierenberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (9):
- United States (9):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Synergy Research Centers, San Diego, California
  - Atlanta Institute of Medicine & Research, Inc., Altanta, Georgia
  - Capital Clinical Research Associates, Rockville, Maryland
  - NorthCoast Clinical Trials, Beachwood, Ohio
  - CRI Worldwide, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 9 study centers between April and December 2008
Groups:
- BCI-024 and BCI-049 (Buspirone and Melatonin): 1 over-encapsulated tablet of buspirone 15 mg and 1 over-encapsulated tablet of melatonin 3 mg QD
- BCI-024 (Buspirone): 1 over-encapsulated tablet of buspirone 15 mg QD
- Placebo: Matching placebo QD
Period: Enrolled
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin) | BCI-024 (Buspirone) | Placebo
Started | 71 | 37 | 34
Completed | 67 | 34 | 33
Not Completed | 4 | 3 | 1
Period: Treated
Arm/Group | BCI-024 and BCI-049 (Buspirone and Melatonin) | BCI-024 (Buspirone) | Placebo
Started | 67 | 34 | 33
Completed | 54 | 28 | 30
Not Completed | 13 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- BCI-024 and BCI-049: Buspirone 15 mg and Melatonin 3 mg QD
- BCI-024: Buspirone 15 mg QD
- Placebo: Placebo QD
- Total: Total of all reporting groups
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo | Total
Number analyzed (Participants) | 67 | 34 | 33 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 34 | 33 | 134
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (12.06) | 40.8 (12.55) | 42.7 (11.62) | 42.4 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 20 | 24 | 87
  Male | 24 | 14 | 9 | 47
Region of Enrollment [Number; unit: participants]
  United States | 67 | 34 | 33 | 134

OUTCOME MEASURES:

1. Primary Outcome: The Score on the Clinical Global Impression-Improvement (CGI-I) at Week 6
Description: Clinical Global Impression (CGI) is a standardized, clinician-rated assessment designed to allow the clinician to rate severity of illness, change over time, and pharmacologic treatment effects with consideration of the patient's clinical condition and the severity of side effects experienced (Guy 1976). Specifically, it consists of two global subscales: Global Improvement (CGI-I) Severity of Illness (CGI-S)
  The CGI-I was administered at Weeks 2, 4 and 6. The CGI-I evaluation was performed with instruction to "Rate the patient's total improvement whether or not, in your judgment, it is due entirely to drug treatment." The Investigator was asked "Compared to the patient's condition at the Baseline visit, please assign a rating to how much the patient changed." Responses for the CGI-I evaluation included the following categories:
  0: Not Assessed
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Week 6
Population: 142 subjects were enrolled and randomized in the study. 8 of these subjects were randomized but never received study drug. Subjects included in the MITT analysis received at least 1 dose of study drug and provided at least 1 post-baseline CGI-I assessment. Subjects included in the analysis of safety received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- BCI-024+BCI-049: Buspirone 15 mg and Melatonin 3 mg QD
Arm/Group | BCI-024+BCI-049 | BCI-024 | Placebo
Number analyzed (Participants) | 67 | 34 | 33
units on a scale | 2.37 (0.97) | 2.82 (1.24) | 2.86 (1.09)

2. Secondary Outcome: The Change From Baseline in the CGI-S at Week 6
Description: Clinical Global Impression (CGI) is a standardized, clinician-rated assessment designed to allow the clinician to rate severity of illness, change over time, and pharmacologic treatment effects with consideration of the patient's clinical condition and the severity of side effects experienced (Guy 1976). The CGI-S is a sub-scale of the Clinical Global Impression. The Investigator was asked: "Considering your total clinical experience with patients with this particular population, please assign a rating to how mentally ill the subject is at this time."
  Possible responses include the following:
  0: Not Assessed
  1. Normal, not ill at all
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients. The change from baseline CGI-S score was calculated as the baseline CGI-S score minus the post-baseline CGI-S score, such that a positive change indicated an improvement from baseline.
Time Frame: Baseline and Week 6
Population: Efficacy analysis were completed for the MITT Population: Subjects included in the MITT analysis received at least 1 dose of study drug and provided at least 1 post-baseline CGI-I assessment. Subjects included in the analysis of safety received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo
Number analyzed (Participants) | 67 | 34 | 33
units on a scale | 1.43 (1.08) | .93 (1.07) | 0.97 (1.16)

3. Secondary Outcome: The Change From Baseline in the IDS-C30 at Week 6
Description: The Inventory of Depressive Symptomatology is a 30-item scale that assesses criteria including mood, concentration, self criticism, suicidal ideation, interest, energy/fatigue, sleep, decrease/increase in appetite or weight, psychomotor agitation or retardation, diurnal mood variation, capacity for pleasure, sexual interest, bodily aches and pains, panic or phobic symptoms, digestive problems, interpersonal rejection sensitivity, and leaden paralysis. Items are scored on a 4 point scale with 0 reflecting no symptoms and 3 reflecting symptoms of maximum severity. The total score is calculated by summing the scores from 28 of the 30 items. Only one of items 11 or 12, and only one of items 13 or 14 are scored. The minimum score is 0 and the maximum score is 84. A score of 84 indicates maximum severity of depressive symptoms. Change from baseline is calculated as the baseline score minus the post-baseline score. A positive change indicates improvement.
Time Frame: Week 0 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo
Number analyzed (Participants) | 67 | 34 | 33
units on a scale | 19.24 (1.60) | 16.35 (2.22) | 14.42 (2.14)

4. Secondary Outcome: The Change From Baseline in the Quick Inventory of Depressive Symptomatology - 16 Item Self-Report (QIDS-SR16) at Week 6
Description: The QIDS-SR16 is a 16 question, patient rated scale that assesses the 9 Diagnostic & Statistical Manual of Mental Disorders-IV-Text Revision criterion diagnostic symptom domains including sad mood, concentration, self criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance, decrease or increase in appetite or weight, & psychomotor agitation or retardation. Each item is measured on a scale of 0 to 3. To find total score, you enter:
  1. highest score from items 1-4 (Sleep Items)
  2. item 5 score
  3. highest score from items 6-9 (appetite/weight)
  4. item 10 score
  5. item 11 score
  6. item 12 score
  7. item 13 score
  8. item 14 score
  9. highest score from items 15-16 (psychomotor) These 9 scores are summed to find total score. Total minimum score is 0 units on a scale & total maximum score is 27 units, where higher scores indicate more severe depression. Change from baseline is calculated as baseline score minus Week 6 score. A positive change indicates improvement
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo
Number analyzed (Participants) | 67 | 34 | 33
units on a scale | 8.57 (0.66) | 6.65 (0.92) | 7.31 (0.89)

5. Secondary Outcome: The Change From Baseline on the HAM-A at Week 6
Description: The 14-item HAM-A scale rates the patient's level of anxiety based on feelings of anxiousness, tension, and depression; any phobias, sleep disturbance, or difficulty in concentrating; the presence of genitourinary, cardiovascular, respiratory, autonomic or somatic symptoms; and the interviewer's assessment of the patient's appearance and behavior during the interview. Each item is to be scored on a 5 point scale with 0 reflecting no symptoms and 4 reflecting symptoms of maximum symptom severity (Hamilton 1960).
  The items are summed to find the total score. The total minimum score is 0 units on a scale and the total maximum score is 56 units on a scale, where higher scores indicate more severe anxiety. Change from baseline is calculated as baseline score minus Week 6 score. A positive change indicates improvement.
Time Frame: Week 0 and Week 6
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo
Number analyzed (Participants) | 67 | 34 | 33
units on a scale | 9.04 (0.87) | 6.69 (1.20) | 6.51 (1.16)

ADVERSE EVENTS:
Arm/Group | BCI-024 and BCI-049 | BCI-024 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 16/67 | 7/34 | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCI-024 and BCI-049 (N=67) | BCI-024 (N=34) | Placebo (N=33)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No